CLINICAL TRIAL: NCT03215745
Title: Trial Randomized, Double-blind, Controlled of Delirium Prevention Program in Patients From the Intensive Care Unit Los Comuneros Hospital University of Bucaramanga, Colombia
Brief Title: Delirium Prevention in Patients From the Intensive Care Unit (DELA)
Acronym: DELA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Santander (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 012-2014
Record Dates: First submitted 2017-07-10; First posted 2017-07-12 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Hypoactive Delirium; Hyperactive Delirium; Delirium of Mixed Origin
Keywords: Delirium; Critical Care; Prevention & control; Clinical Trial
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delirium prevention program (Experimental): Delirium prevention program involved a non-pharmacologic preventive interventions that will be focused in: Delirium prevention program includes individualized non-pharmacological interventions such as multisensory stimulation, cognitive stimulation, activate the functional and family involvement.
  Interventions: Behavioral: Delirium prevention program
- Control group (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Delirium prevention program — Delirium prevention program Placard with the names of the care team and the calendar days; cognitively stimulating activities three times a day. Pictures, radio, robe. Visual aids large print books, with daily reinforcement of use Maintain adequate lighting opening blinds and curtains during the day, and darken their environment at night. Dissipation wax and special techniques of communication, with daily reinforcement of these adaptations. Go to the patient by name and tone of voice appropriate. Always listen. Use simple and clear language, face-to-face. Avoid excessive familiarity and childish. Promote family involvement in self-care and caregivers and the reorientation of the patient, contact with extended family during the stay.
  Arms: Delirium prevention program

SUMMARY:
"To determine the efficacy of program of prevention of delirium in critically ill patients from the intensive care units of Bucaramanga and Floridablanca. Methods: The study will be a randomized controlled clinical trial in 600 critically ill patients recruited at 24 hours from arrival on the intensive care units of Bucaramanga and Floridablanca, without delirium, with ≥50% in the PREDELIRIC scale score, who comply with the inclusion and exclusion. The patients will be randomized in blocks to one of the two groups, intervention group (delirium prevention program, n=200) with control group (usual care; n= 400), the study will compare the incidence of delirium in both groups. Patients will be followed every day with Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) until the patient presents delirium, exit to hospitalization or death. Delirium prevention program includes individualized nonpharmacological interventions such as multisensory stimulation, cognitive stimulation, activate the functional and family involvement. The study has received ethical approval from the University of Santander"

DETAILED DESCRIPTION:
"delirium predominance in the intensive care unit (ICU) is 20- 80%, depending on the scale to which it measures itself and some characteristics of the patients ( Carrillo & Sosa, 2010). The development of the delirium in the intensive care unit presents an important impact in the treatment of the patient , therefore directly influences the hospital cost , in the stay and the mortality .Martinez & others (2004) also , the delirium is diagnosed just in 66-84% of the patients who present this complication , because in come circumstances it is confused with dementia or anxiety and why there does not exist a diagnostic methodology adequate for its evaluation. With regard to the diagnosis of the delirium , several methods exist for the diagnosis , the evaluation method of the confusion CAMICU of the english confusion assesment method for the ICU is the most used, in the intensive care unit , for its high sensibility, reliability and validity to identify delirium when it is used by nurses and doctors of the ICU and only it needs 2-3 minutes for its achievement (Ely & others, 2004) This way, Boogaard and collaborators decided to construct and validate a model who allows to predict the delirium probability in adult patients of intensive care unit (Boogaard

* others, 2012), in order to restore preventive measurements to reduce its incidence, gravity and duration. The delirium have high frequency and with an impact bio-psico-economic in the patient and its environment , the prevention is the most effective and economic measure of tackling the delirium in its initial phase and nursing contributes to a great extent in this work . It is as well as in a titled previous study : validity of the model of prediction of the delirium in intensive care unit of Bucaramanga, realized by Torres and Páez in 2014 in the Comuneros universitarian Hospital of Bucaramanga brought up to the date an incidence of the delirium of 20.5%, with a mortality of 47.5% of the patients who do delirium during its stay in ICU , proving the efficacy od the model PREDELIRIC to predict the delirium in the first 24 hours of stay in ICU , in patients with high values its like say a PREDELIRIC result >50% Taking this study as a precedent there appears the target to determine the efficacy of the prevention program of delirium in the population of critical patients in Bucaramanga, (the Comuneros universitarian Hospital of Bucaramanga) across a randomized controlled clinical essay , in order to predict early in these patients the possibility of delirium development and to facilitate the application of preventive measurements not pharmacological in patients with high risk . these preventive measurements would be done across individualized interventions and they would be focused after the improved orientation , cognitive stimulation , early mobilization to listen to music with the intention of reduce the delirium incidence, of improving the cognition of the patients and avoiding its deterioration during the staying in the ICU , condition that can remain after its departure ( Inouye & others, 1999). Also, the results of this investigation will appear in a scientific article and scientific congresses in the área of health . Also, they will be announced to the universitarian community and the involved institution. Key words : Delirium, intensive care, prevention , nursing interventions. Like an important antecedent in Santander the group of research of the nursing program Everest execute a study to validate the prediction model PREDELIRIC to a spanish version , this study expose the need to identify and implement interventions of nursing to prevent the delirium in critical patients of Bucaramanga Our priority now is to apply the model of prediction PREDELIRIC validated in a spanish version to the population of critical patients to predict early in these patients the possibility of development of delirium , facilitating the specific application of not pharmacological preventive measurements in patient who is in high risk. These preventive measurements would be done across an individualized intervention and they would be focused to: to improve the orientation, cognitive stimulation , early mobilization, listen to music, in patients of high risk, Inouye & others (1999) All this , focused to improve the cognition of the patients and to avoid the cognitive deterioration presented during the stay in the ICU and that can remain after the departure of the patient in the ICU, Inouye
* others (1999) Additionally identifying in a specific way the patients who has a benefit from the preventive measurements optimizes the time of personnel of health, reducing the incidence of the delirium, turns into a strategy cost- benefit for the persons and the relatives also for the institution on having diminished the hospitable stay, adverse events and the morbi- mortality . Inouye & others (1990). It is of clarifying and admitting that now some institutions make different interventions, which tackle the prevention of the delirium, however , these interventions are realized in an isolated way, associated with the interest and motivation of the personnel, there do not exist organized and systematized processes that they allow to face and link to the whole personnel , the recognition of the delirium during the hospitalization in the ICU , and although they interfere in the process , there do no exist very few concrete proposals that reflect in wich way institutions impact the presentation and prevention of the delirium . In the same way , the services of intensive care unit has been unidentified that the recommendations with regard to the care and prevention of the delirium tend yo be generalized, without dedicating enough time to the recognition of the problems, neither is clear the process of pursuit that is done, to the needs and to the result of the realized interventions . To the date conclusive studies are not known in this subject and there has not been proved the efficacy of not pharmacological interventions directed to the prevention of the delirium in critics patients, only there exist the modality of the study of doctor Inouye and collaborators in 1999 who verified a decrease of 30% of the delirium with the implementation of these measurements in hospitalized aged patients. Inouye & others (1999) Bearing in mind the serious and irreversible consequences of the delirium to shortly and long term in the critical patients, we want to propose the implementation of not pharmacological measurements to prepare this phenomenon and simultaneously to prove the efficacy in patients that diagnoses a high risk of development of delirium as the application of the scale PREDELIRIC version validated in spanish The investigation on the prediction of the delirium , of indirect form will tackle these problematic , generating knowledge on the real e situation, favoring the identification of courses that will face processes, qualification of the personnel and making of a guide of intervention in nursing focus on the diminish the frenzy of the intensive unit care of the country One admits that beyond the requested for the regulations , the training and permanent accompaniment is needed for the team of health as regards the attention humanized in highly specializing and technological stages as it is the ICU To obtain new knowledge that they can contribute to the comprehension and the sensitization of the situation of the delirium in the persons hospitalized in the intensive care unit does part of the contribution to the body of knowledge in the área of critical care , it is so to find a predictor of the investigation of delirium cost in the intensive care unit strengthens the theoretical bases to improve the care . There will be beneficiaries of the results of the present investigation, in addition to the patients , relatives and personnel of health, the educational institutions of the region , who will have new indications to the academic programs realizing on the programs of specialization of the área, this way to validate the care interventions for the user who came to the ICU and improve the offered care. Generating and applying the results of the present study will be a contribution for the generation of models of attention in Colombia, directed to a persons who live through an illness situation and who are hospitalized in ICU , thinking about hoe to high light the importance of implementing strategies for the advance in the knowledge and the employment of the results in the formation, practice and investigation to consolidate the proposals to answer for the needs of this population . The results of the present study will be presented like a proposal for the institutions and specially for the intensive care unit adult with the target to offer tools to the care, this will be a progress of the general satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Be older than 18 years
* To have 24 hours of stay from the ingress to the intensive care unit
* To expire with the criteria of intensive care unit defined by the investigative group (it presents itself with support, with invasive mechanical ventilation.
* Patient without delirium in the revenue
* Patients who present a percentage of prediction bigger than 50% according to the model PREDELIRIC

Exclusion Criteria:

* Patients who scale of sedation RASS is applied and have like result of +4 and +5( scale that is applied systematically to the patient in intensive care unit)
* Subjects with cognitive deficit or previous mental illness
* Patients with precedents previous to delirium or in which the delirium measurement could be affected by its base condition
* Patients with alcoholism precedents.
* To be at the moment of the application of the instruments under substances that limit its skill to communicate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Delirium | Within the first 30 days after admission at ICW
  For the measurement of delirium will be with the instrument Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) version in spanish.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia C Torres, RN, MSc, Principal Investigator — Universidad de Santander
Locations (1):
- Los Comuneros Hospital University of Bucaramanga, Bucaramanga, Santander Department, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Contreras CCT, Esteban ANP, Parra MD, Romero MKR, Silva CGD, Buitrago NPD. Multicomponent nursing program to prevent delirium in critically ill patients: a randomized clinical trial. Rev Gaucha Enferm. 2021 Nov 3;42:e20200278. doi: 10.1590/1983-1447.2021.20200278. eCollection 2021. English, Spanish. PMID 34755800